CLINICAL TRIAL: NCT04540315
Title: Reducing Surgical Readmissions Through Mobile Technology: A Randomized Controlled Trial
Brief Title: Reducing Surgical Readmissions Through Mobile Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-0739; MSN225549 (Other Grant/Funding Number: ASSOCIATION FOR VA SURGEONS); A539722 (Other: University of Wisconsin, Madison); SMPH/SURGERY (Other: University of Wisconsin, Madison); Protocol Version 9/20/2021 (Other: UW Madison)
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Readmission; Perioperative Care
Keywords: mobile app; readmission

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - MobiMD app (Experimental): Intervention group will receive notifications to their smart device through MobiMD app. Participants will be asked to fill out reports and upload all clinically relevant data using the app. Engaging with the app will be in addition to the standard of care follow-up.
  Interventions: Behavioral: MobiMD
- Standard of Care (No Intervention): The standard of care control group will receive conventional postoperative care. Participants will receive reported outcome survey by email.

INTERVENTIONS:
Behavioral: MobiMD — MobiMD is a mobile app. This is an app available to IOS and Android devices only. The app provides a digitized version of the discharge instructions and provides push notifications to remind the participant of important instructions. In addition, the app allows participants (and their care teams) to record and track relevant clinical data.
  Arms: Intervention - MobiMD app

SUMMARY:
This randomized trial will study the effect of a mobile app that facilitates patient engagement (patients undergoing complex abdominal surgery will track metrics of interest to the surgeon, submit reports on their symptoms/pain/physical function, and upload wound images) on readmission to the hospital. This trial will also assess whether the app can impact surgical complication severity, number of emergency department visits, and readmission costs. 300 participants will be enrolled and can expect to be on study for 6 months.

DETAILED DESCRIPTION:
Hospital readmissions are estimated to cost $17.4 billion per year in the Medicare population alone. Readmission rates may be as high as 30% for patients undergoing complex abdominal surgery. In this study, investigators will conduct a randomized controlled trial (RCT) to assess the effect of a novel mobile technology platform, MobiMD, on hospital readmission in complex abdominal surgery patients. Data from a 50-patient MobiMD pilot study supports the RCT design and mobile platform's feasibility in this study population. Investigators hypothesize that the MobiMD app can facilitate better information transfer between surgeons and patients in the high-risk postoperative time period, thereby reducing hospital readmissions, emergency department visits, complication severity, and overall resource utilization.

Investigators will conduct a parallel, single-blinded, 2-arm randomized controlled trial investigating the effect of a novel mobile health app on hospital readmissions for adults undergoing complex abdominal surgery. Three hundred participants (150 patients per arm) will be randomized to compare standard postoperative care alone versus plus MobiMD app. This study is powered to detect a clinically meaningful difference of 11% in readmissions. Participants will be eligible if they undergo any of the following procedures: pancreaticoduodenectomy, cytoreductive surgery/ hyperthermic intraperitoneal chemotherapy (HIPEC), gastrectomy, distal pancreatectomy, liver transplant, pancreas transplant, simultaneous kidney and pancreas transplant, low anterior resection, and any bowel resection requiring an ostomy. The MobiMD app collects important clinical data points and patient-reported outcomes with associated push notifications sent directly to the patient's smart device. Clinical data collected via the MobiMD app include vital signs, red flag symptoms, daily wound and surgical drain images, ostomy output, drain output, medication compliance, and wound care compliance.

The primary outcome of the RCT will be 30-day hospital readmission. The secondary outcomes will include 90-day readmission, emergency department and urgent care visits, complication severity, and total readmission cost. Exploratory outcomes will include length of stay and patient-reported outcomes in patient satisfaction, pain, and physical function. All participants will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* English speaking
* Able to pass a cognitive screening test
* Patient or caregiver has access to a device capable of running the MobiMD app (tablet or smartphone).
* Undergoing complex abdominal surgery in the departments of surgical oncology, colorectal surgery, or transplant surgery, (Complex abdominal surgery is interpreted as whipple procedure, hyperthermic intraperitoneal chemotherapy (HIPEC), gastrectomy, distal pancreatectomy, liver transplant, pancreas transplant, simultaneous kidney and pancreas transplant, low anterior resection, and all bowel resections requiring an ostomy).

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Proportion of participants readmitted within 30 days of surgery | 30 days postoperative
  The primary aim of the study is to determine if using MobiMD app changes the proportion of participants readmitted to the hospital within 30 days of surgery. Readmission will be counted as "1" event and no readmission will be counted as "0" event. In concordance with the standards of Centers for Medicare and Medicaid services, multiple readmissions for the same participant within a 30-day period will be measured as one event.

SECONDARY OUTCOMES:
Proportion of participants readmitted within 90 days of surgery | 90 days post-operative
  Readmission will be counted as "1" event and no readmission will be counted as "0" event. In concordance with the standards of Centers for Medicare and Medicaid services, multiple readmissions for the same participant within a 90-day period will be measured as one event.
30 day postoperative complication severity as measured by Clavien-Dindo Score | 30 days postoperative
  Complications and their associated severity as measured by the Clavien-Dindo score will be reported at 30 days postoperatively. The Clavien-Dindo score ranges from 1 to 5, with higher score indicating more severe complication. This score will be obtained and scored from chart review.
90 day postoperative complication severity as measured by Clavien-Dindo Score | 90 days postoperative
  Complications and their associated severity as measured by the Clavien-Dindo score will be reported at 90 days postoperatively. The Clavien-Dindo score ranges from 1 to 5, with higher score indicating more severe complication. This score will be obtained and scored from chart review.
Total number of emergency department visits at 30 days postoperative | 30 days postoperative
  The total number of emergency department and urgent care visits will be reported at 30 days postoperatively. This data will be obtained from chart review.
Total number of emergency department visits at 90 days postoperative | 90 days postoperative
  The total number of emergency department and urgent care visits will be reported at 90 days postoperatively. This data will be obtained from chart review.
Total readmission cost | Up to 90 days postoperative
  The total readmission hospital cost will be calculated using fiscal data harvested form Clarity (Epic). Clarity includes direct/indirect and fixed/variable hospital cost and reimbursement for professional fees. These variables can be accessed in very short timeframes (1 week). The two trial arms will be compared with respect to total healthcare-associated readmission costs.

OTHER OUTCOMES:
30-day participant satisfaction measured by Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey | 30 days postoperative
  Participant satisfaction will be measured at 30 days using the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey. The CAHPS Surgical Care (S-CAHPS) survey focuses on key areas of perioperative patient care, including preoperative, day of operation, and postoperative care. As study intervention focuses on postoperative care, participants will be supplied with the portion of the questionnaire related to postoperative care (questions 26-35).
90-day participant satisfaction measured by Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey | 90 days postoperative
  Participant satisfaction will be measured at 90 days using the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey. The CAHPS Surgical Care (S-CAHPS) survey focuses on key areas of perioperative patient care, including preoperative, day of operation, and postoperative care. As study intervention focuses on postoperative care, participants will be supplied with the portion of the questionnaire related to postoperative care (questions 26-35).
180-day participant satisfaction measured by Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey | 180 days postoperative
  Participant satisfaction will be measured at 180 days using the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey. The CAHPS Surgical Care (S-CAHPS) survey focuses on key areas of perioperative patient care, including preoperative, day of operation, and postoperative care. As study intervention focuses on postoperative care, participants will be supplied with the portion of the questionnaire related to postoperative care (questions 26-35).
30-day physical function as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) short form score | 30 days postoperative
  Patient-reported outcomes in physical function will be collected at 30-days post-operatively. The outcome measure will be assessed by the NIH PROMIS short forms, which can be administered through the MobiMD app. The PROMIS Short Forms will be used and are publicly available from healthmeasures.net.
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life. The functional performance tests assess physical abilities (strength, mobility) in ways that are relevant to daily living. The short form consists of questions which can be answered on a scale of 1-5, where 1-unable to do, 2-with much difficulty, 3-with some difficulty,4-with a little difficulty, 5- without any difficulty. A higher scores correlates to more physically active person.
90-day physical function as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) short form score | 90 days postoperative
  Patient-reported outcomes in physical function will be collected at 90-days post-operatively. The outcome measure will be assessed by the NIH PROMIS short forms, which can be administered through the MobiMD app. The PROMIS Short Forms will be used and are publicly available from healthmeasures.net.
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life. The functional performance tests assess physical abilities (strength, mobility) in ways that are relevant to daily living. The short form consists of questions which can be answered on a scale of 1-5, where 1-unable to do, 2-with much difficulty, 3-with some difficulty,4-with a little difficulty, 5- without any difficulty. A higher scores correlates to more physically active person.
180-day physical function as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) short form score | 180 days postoperative
  Patient-reported outcomes in physical function will be collected at 180-days post-operatively. The outcome measure will be assessed by the NIH PROMIS short forms, which can be administered through the MobiMD app. The PROMIS Short Forms will be used and are publicly available from healthmeasures.net.
  The PROMIS short forms are self-report instruments used to measure aspects of quality of life. The functional performance tests assess physical abilities (strength, mobility) in ways that are relevant to daily living. The short form consists of questions which can be answered on a scale of 1-5, where 1-unable to do, 2-with much difficulty, 3-with some difficulty,4-with a little difficulty, 5- without any difficulty. A higher scores correlates to more physically active person.
30-day pain intensity as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) short form pain intensity scale | 30 days postoperative
  Patient-reported outcomes in physical function will be collected at 30-days post-operatively. The outcome measure will be assessed by the NIH PROMIS short forms, which can be administered through the MobiMD app. The PROMIS Short Form v2.0 - Pain Intensity measure will be used and is publicly available from healthmeasures.net.
  PROMIS pain intensity scale consists of 3 questions which can be answered on a scale of 1-5, where 1- had no pain, 2- mild pain, 3- moderate pain, 4- severe pain, 5- very severe pain. The cumulative score can range from 5-15, where higher scores correlates to more pain.
90-day pain intensity as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) short form pain intensity scale | 90 days postoperative
  Patient-reported outcomes in physical function will be collected at 90-days post-operatively. The outcome measure will be assessed by the NIH PROMIS short forms, which can be administered through the MobiMD app. The PROMIS Short Form v2.0 - Pain Intensity measure will be used and is publicly available from healthmeasures.net.
  PROMIS pain intensity scale consists of 3 questions which can be answered on a scale of 1-5, where 1- had no pain, 2- mild pain, 3- moderate pain, 4- severe pain, 5- very severe pain. The cumulative score can range from 5-15, where higher scores correlates to more pain.
180-day pain intensity as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) short form pain intensity scale | 180 days postoperative
  Patient-reported outcomes in physical function will be collected at 180-days post-operatively. The outcome measure will be assessed by the NIH PROMIS short forms, which can be administered through the MobiMD app. The PROMIS Short Form v2.0 - Pain Intensity measure will be used and is publicly available from healthmeasures.net.
  PROMIS pain intensity scale consists of 3 questions which can be answered on a scale of 1-5, where 1- had no pain, 2- mild pain, 3- moderate pain, 4- severe pain, 5- very severe pain. The cumulative score can range from 5-15, where higher scores correlates to more pain.
Total number of days spent in-hospital for the readmission event | Up to 90 days
  Readmission length of stay will be measured as the total number of days spent in-hospital for the readmission event. This data will be obtained from chart review and will include date of readmission through date of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I Voils, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diehl TM, Barrett JR, Abbott DE, Cherney Stafford LM, Hanlon BM, Yang Q, Van Doorn R, Weber SM, Voils CI. Protocol for the MobiMD trial: A randomized controlled trial to evaluate the effect of a self-monitoring mobile app on hospital readmissions for complex surgical patients. Contemp Clin Trials. 2022 Feb;113:106658. doi: 10.1016/j.cct.2021.106658. Epub 2021 Dec 22. PMID 34954099